CLINICAL TRIAL: NCT03780335
Title: EARLY Microvascular Dysfunction Prediction Using Quantitative Flow Ratio After ST-segment Elevation MYOcardial Infarction (EARLY-MYO-QFR I)
Brief Title: Early Prediction of QFR in STEMI-I
Acronym: EARLYmyo-QFR-I
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 16CR3034A
Record Dates: First submitted 2018-12-10; First posted 2018-12-19 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2018-08

CONDITIONS: ST Segment Elevation Myocardial Infarction
Keywords: STEMI; Cardiac magnetic resonance
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MVO group: CMR was performed in all the cases. According to the results of CMR, we divided the study population into MVO group and Non-MVO group.
  Interventions: Diagnostic Test: Computation of quantitative flow ratio
- Non-MVO group: CMR was performed in all the cases. According to the results of CMR, we divided the study population into MVO group and Non-MVO group.
  Interventions: Diagnostic Test: Computation of quantitative flow ratio

INTERVENTIONS:
Diagnostic Test: Computation of quantitative flow ratio — Computation of QFR was performed offline, using AngioPlus system(Pluse medical imaging technology, Shanghai, China). In the first step, 2 diagnostic angiographic projections before PCI, at least 25° apart, were selected and 3D reconstruction of the interrogated vessel without its side branches was performed. Then, the software computed the QFR.

SUMMARY:
The study intends to provide important data on whether the noval method using quantitative flow ratio could predict microvascular dysfunction.

DETAILED DESCRIPTION:
Microvascular dysfunction (MVD) is a serious complication of PCI, which happens frequently after STEMI and always correlates with a poor prognosis. However, precise and simplified assessment of MVD is difficult, especially in the acute phase of STEMI patients. Resent studies suggested that FFR could be overestimated when MVD exists. But whether the overestimated value of FFR caused by CMR defined MVO could reflect microcirculation function is still unclear.

This study is a retrospective study using STEMI patients with TFG 2/3 of the infarct vessel on initial angiography and presumed culprit lesion ≥50% as the population. Contrast-enhanced CMR was performed 5 days after PCI as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients treated with revasculation within 12 hours from onset of symptoms to PCI time and received CMR 5 days afterwards. STEMI was defined as a combination of the following: chest pain for more than 30min, electrocardiographic (ECG) changing with ST segment elevation of >2 mm in at least 2 precordial leads and >1 mm in limb leads, and abnormal troponin levels or CKMB levels higher than twice the upper limit of normal.
* Patients with TFG 2/3 in the initial angiography of the culprit vessel.

Exclusion Criteria:

* Patients with left bundle branch block in the presenting ECG, cardiogenic shock, PCI or bypass surgery history.
* Patients with residual stenosis <50%.
* Patients with unqualified coronary angiographic images with problems such as ostial lesion, severe vessel tortuosity and diffuse long lesions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: STEMI patients who underwent successful reperfusion therapy with TFG 2/3 of the infarct vessel on initial angiography and presumed culprit lesion ≥50%.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Cardiac magnetic resonance (CMR) | Five days after PCI
  Cardiac magnetic resonance (CMR) is a non-invasive test for MVO assessing

SECONDARY OUTCOMES:
TIMI Flow Grade (TFG) | One mins before PCI
  TIMI Flow Grade (TFG) assesses flow in the epicardial arteries. Type zero perfusion expressed not antegrade movement away the occlusion; type two is a minimum, inadequate perfusion of contrast average round the mass; type three (partial perfusion) is a perfect just limited perfusion from the distal coronary bed by contrast element; and type three (complete perfusion) is an antegrade movement to the whole distal artery at a regular flow.
TIMI Flow Grade (TFG) | One mins after PCI
  TIMI Flow Grade (TFG) assesses flow in the epicardial arteries. Type zero perfusion expressed not antegrade movement away the occlusion; type two is a minimum, inadequate perfusion of contrast average round the mass; type three (partial perfusion) is a perfect just limited perfusion from the distal coronary bed by contrast element; and type three (complete perfusion) is an antegrade movement to the whole distal artery at a regular flow.
TIMI Myocardial Perfusion Grade (TMPG) | One mins before PCI
  TIMI Myocardial Perfusion Grade (TMPG) assesses flow in the micrevessels. TMPG0: no or minimal blush; TMPG1: Stain present Blush persists on next injection; TMPG2: Dye strongly persistent at end of washout Gone by next injection; TMPG3: normal ground glass appearance of blush Dye mildly persistentat end of washout.
TIMI Myocardial Perfusion Grade (TMPG) | One mins after PCI
  TIMI Myocardial Perfusion Grade (TMPG) assesses flow in the micrevessels. TMPG0: no or minimal blush; TMPG1: Stain present Blush persists on next injection; TMPG2: Dye strongly persistent at end of washout Gone by next injection; TMPG3: normal ground glass appearance of blush Dye mildly persistentat end of washout.

REFERENCES:
- [Background] Niccoli G, Burzotta F, Galiuto L, Crea F. Myocardial no-reflow in humans. J Am Coll Cardiol. 2009 Jul 21;54(4):281-92. doi: 10.1016/j.jacc.2009.03.054. PMID 19608025
- [Background] Sheng X, Ding S, Ge H, Sun Y, Kong L, He J, Pu J, He B. Intracoronary infusion of alprostadil and nitroglycerin with targeted perfusion microcatheter in STEMI patients with coronary slow flow phenomenon. Int J Cardiol. 2018 Aug 15;265:6-11. doi: 10.1016/j.ijcard.2018.04.119. Epub 2018 Apr 25. PMID 29728334
- [Background] Fearon WF, Balsam LB, Farouque HM, Caffarelli AD, Robbins RC, Fitzgerald PJ, Yock PG, Yeung AC. Novel index for invasively assessing the coronary microcirculation. Circulation. 2003 Jul 1;107(25):3129-32. doi: 10.1161/01.CIR.0000080700.98607.D1. Epub 2003 Jun 23. PMID 12821539
- [Background] Fearon WF, Shah M, Ng M, Brinton T, Wilson A, Tremmel JA, Schnittger I, Lee DP, Vagelos RH, Fitzgerald PJ, Yock PG, Yeung AC. Predictive value of the index of microcirculatory resistance in patients with ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2008 Feb 5;51(5):560-5. doi: 10.1016/j.jacc.2007.08.062. PMID 18237685
- [Background] Fearon WF, Low AF, Yong AC, McGeoch R, Berry C, Shah MG, Ho M, Kim HS, Loh JP, Oldroyd KG. Response to letter regarding article, "Prognostic value of the index of microcirculatory resistance measured after primary percutaneous coronary intervention". Circulation. 2014 Feb 18;129(7):e342. doi: 10.1161/CIRCULATIONAHA.113.007271. No abstract available. PMID 24550557
- [Background] van de Hoef TP, Nolte F, EchavarrIa-Pinto M, van Lavieren MA, Damman P, Chamuleau SA, Voskuil M, Verberne HJ, Henriques JP, van Eck-Smit BL, Koch KT, de Winter RJ, Spaan JA, Siebes M, Tijssen JG, Meuwissen M, Piek JJ. Impact of hyperaemic microvascular resistance on fractional flow reserve measurements in patients with stable coronary artery disease: insights from combined stenosis and microvascular resistance assessment. Heart. 2014 Jun;100(12):951-9. doi: 10.1136/heartjnl-2013-305124. Epub 2014 Apr 11. PMID 24727867
- [Background] Tu S, Echavarria-Pinto M, von Birgelen C, Holm NR, Pyxaras SA, Kumsars I, Lam MK, Valkenburg I, Toth GG, Li Y, Escaned J, Wijns W, Reiber JH. Fractional flow reserve and coronary bifurcation anatomy: a novel quantitative model to assess and report the stenosis severity of bifurcation lesions. JACC Cardiovasc Interv. 2015 Apr 20;8(4):564-74. doi: 10.1016/j.jcin.2014.12.232. Epub 2015 Mar 26. PMID 25819180
- [Background] Emori H, Kubo T, Kameyama T, Ino Y, Matsuo Y, Kitabata H, Terada K, Katayama Y, Aoki H, Taruya A, Shimamura K, Ota S, Tanaka A, Hozumi T, Akasaka T. Diagnostic Accuracy of Quantitative Flow Ratio for Assessing Myocardial Ischemia in Prior Myocardial Infarction. Circ J. 2018 Feb 23;82(3):807-814. doi: 10.1253/circj.CJ-17-0949. Epub 2018 Jan 16. PMID 29343675
- [Background] Spitaleri G, Tebaldi M, Biscaglia S, Westra J, Brugaletta S, Erriquez A, Passarini G, Brieda A, Leone AM, Picchi A, Ielasi A, Girolamo DD, Trani C, Ferrari R, Reiber JHC, Valgimigli M, Sabate M, Campo G. Quantitative Flow Ratio Identifies Nonculprit Coronary Lesions Requiring Revascularization in Patients With ST-Segment-Elevation Myocardial Infarction and Multivessel Disease. Circ Cardiovasc Interv. 2018 Feb;11(2):e006023. doi: 10.1161/CIRCINTERVENTIONS.117.006023. PMID 29449325
- [Background] Tu S, Westra J, Yang J, von Birgelen C, Ferrara A, Pellicano M, Nef H, Tebaldi M, Murasato Y, Lansky A, Barbato E, van der Heijden LC, Reiber JHC, Holm NR, Wijns W; FAVOR Pilot Trial Study Group. Diagnostic Accuracy of Fast Computational Approaches to Derive Fractional Flow Reserve From Diagnostic Coronary Angiography: The International Multicenter FAVOR Pilot Study. JACC Cardiovasc Interv. 2016 Oct 10;9(19):2024-2035. doi: 10.1016/j.jcin.2016.07.013. PMID 27712739
- [Background] Pu J, Ding S, Ge H, Han Y, Guo J, Lin R, Su X, Zhang H, Chen L, He B; EARLY-MYO Investigators. Efficacy and Safety of a Pharmaco-Invasive Strategy With Half-Dose Alteplase Versus Primary Angioplasty in ST-Segment-Elevation Myocardial Infarction: EARLY-MYO Trial (Early Routine Catheterization After Alteplase Fibrinolysis Versus Primary PCI in Acute ST-Segment-Elevation Myocardial Infarction). Circulation. 2017 Oct 17;136(16):1462-1473. doi: 10.1161/CIRCULATIONAHA.117.030582. Epub 2017 Aug 27. PMID 28844990
- [Background] Cuculi F, De Maria GL, Meier P, Dall'Armellina E, de Caterina AR, Channon KM, Prendergast BD, Choudhury RP, Forfar JC, Kharbanda RK, Banning AP. Impact of microvascular obstruction on the assessment of coronary flow reserve, index of microcirculatory resistance, and fractional flow reserve after ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2014 Nov 4;64(18):1894-904. doi: 10.1016/j.jacc.2014.07.987. Epub 2014 Oct 27. PMID 25444143
- [Background] Mejia-Renteria H, Lee JM, Lauri F, van der Hoeven NW, de Waard GA, Macaya F, Perez-Vizcayno MJ, Gonzalo N, Jimenez-Quevedo P, Nombela-Franco L, Salinas P, Nunez-Gil I, Del Trigo M, Goto S, Lee HJ, Liontou C, Fernandez-Ortiz A, Macaya C, van Royen N, Koo BK, Escaned J. Influence of Microcirculatory Dysfunction on Angiography-Based Functional Assessment of Coronary Stenoses. JACC Cardiovasc Interv. 2018 Apr 23;11(8):741-753. doi: 10.1016/j.jcin.2018.02.014. PMID 29673505
- [Derived] Sheng X, Qiao Z, Ge H, Sun J, He J, Li Z, Ding S, Pu J. Novel application of quantitative flow ratio for predicting microvascular dysfunction after ST-segment-elevation myocardial infarction. Catheter Cardiovasc Interv. 2020 Feb;95 Suppl 1:624-632. doi: 10.1002/ccd.28718. Epub 2020 Jan 8. PMID 31912991